CLINICAL TRIAL: NCT01740310
Title: Vaccine Acceptance in Pregnant Minority Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Saad B. Omer, PhD, Associate Professor, Emory University
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: IRB00057339
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Pregnancy
Keywords: pregnancy,; vaccine acceptance,; vaccination,; influenza,; pertussis,; Tdap,; minority,; African-American
MeSH Terms: conditions — Influenza, Human; Whooping Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Elaboration Video Arm (Experimental): Women randomized to this arm will be exposed to a handheld/electronic tablet device-based video with detailed vaccine-related information designed to invoke a high level of attention to the message and thought (elaboration) while processing information.
  Interventions: Behavioral: Maternal Vaccine Education
- High Elaboration Interactive Tutorial Arm (Experimental): Women will be exposed to a handheld/electronic tablet device-based intervention designed to invoke a high level of attention to the message and thought (elaboration) while processing information through an interactive question/answer format.
  Interventions: Behavioral: Maternal Vaccine Education
- Low Elaboration / Control Arm (Placebo Comparator): Women randomized to the control arm will be provided standard CDC vaccine information statements that will likely lead to low elaboration information processing.
  Interventions: Behavioral: Maternal Vaccine Education

INTERVENTIONS:
Behavioral: Maternal Vaccine Education — It is assumed that the women will also receive vaccine education materials from the OB/GYN practices as part of routine care. The intervention for all three arms will be conducted during routine prenatal office visits. Participants will complete a baseline questionnaire to assess attitudes regarding vaccination and will then be randomized to one of three enrollment arms and will be exposed to an intervention designed to take no longer than 20 minutes, so that patients can complete it during the time they are waiting to be seen. While participants are completing the handheld/electronic tablet device-based intervention, the study recruiter will observe them and document dose exposure to the messages being presented. The enrolled women will be contacted a month after the expected date of delivery and a follow up interview will be conducted to ascertain their vaccination status for receipt of influenza vaccine in pregnancy and Tdap during pregnancy or immediately post-partum.

SUMMARY:
The purpose of study will be to test two vaccine education strategies to learn how they impact flu and pertussis (Tdap) vaccination rates and attitudes regarding vaccination during pregnancy after participating in the intervention. The education strategies will be based on the elaboration likelihood model (ELM). This model is based on experimental psychology and has been previously used to increase breast cancer screening rates. These education strategies will be delivered through routine prenatal care visits to black/African-American women in Atlanta.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant, expecting delivery between August 31, 2012 and June 30, 2013
* Between the ages of 18-50 years old
* Black/African American

Exclusion Criteria:

* Have received the influenza or Tdap vaccine during the current pregnancy
* Already enrolled in the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Influenza vaccination rates in pregnancy | Baseline and one month after participant's expected date of delivery
  Data on vaccination status will be collected from participants enrolled in the main phase of the study during follow up starting one month after the expected date of delivery. We will contact healthcare providers to obtain vaccination records for those who provide written consent to release their immunization records.

SECONDARY OUTCOMES:
Tdap vaccination rates in pregnancy | Baseline and one month after participant's expected date of delivery
  Data on vaccination status will be collected from participants enrolled in the main phase of the study during follow up starting one month after the expected date of delivery. We will contact healthcare providers to obtain vaccination records for those who provide written consent to release their immunization records.
Change in attitudes regarding vaccination | Baseline and one month after the expected date of delivery
  Data on attitudes regarding vaccination status will be collected from participants enrolled in the main phase of the study during follow up starting one month after the expected date of delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Saad B Omer, PhD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Dourron OB/Gyn Associates Clinic, Decatur, Georgia
  - New Millenium Obstetrics & Gynecology, Riverdale, Georgia

REFERENCES:
- [Background] Gust D, Brown C, Sheedy K, Hibbs B, Weaver D, Nowak G. Immunization attitudes and beliefs among parents: beyond a dichotomous perspective. Am J Health Behav. 2005 Jan-Feb;29(1):81-92. doi: 10.5993/ajhb.29.1.7. PMID 15604052
- [Background] Gust DA, Kennedy A, Wolfe S, Sheedy K, Nguyen C, Campbell S. Developing tailored immunization materials for concerned mothers. Health Educ Res. 2008 Jun;23(3):499-511. doi: 10.1093/her/cym065. Epub 2007 Oct 23. PMID 17959583
- [Background] Paulussen TG, Hoekstra F, Lanting CI, Buijs GB, Hirasing RA. Determinants of Dutch parents' decisions to vaccinate their child. Vaccine. 2006 Jan 30;24(5):644-51. doi: 10.1016/j.vaccine.2005.08.053. Epub 2005 Aug 26. PMID 16157423
- [Background] Wilson BJ. Designing media messages about health and nutrition: what strategies are most effective? J Nutr Educ Behav. 2007 Mar-Apr;39(2 Suppl):S13-9. doi: 10.1016/j.jneb.2006.09.001. PMID 17336800
- [Background] Baxter CE, Barata PC. The paradox of HPV vaccines: how to reach sexually inexperienced women for protection against a sexually transmitted infection. Womens Health Issues. 2011 May-Jun;21(3):239-45. doi: 10.1016/j.whi.2010.11.007. Epub 2011 Feb 18. PMID 21330153
- [Background] Petty R, Cacioppo J. Communication and Persuasion: Central and Peripheral Routes to Attitude Change. New York, NY: Springer-Verlag; 1986.
- [Background] Vannice KS, Salmon DA, Shui I, Omer SB, Kissner J, Edwards KM, Sparks R, Dekker CL, Klein NP, Gust DA. Attitudes and beliefs of parents concerned about vaccines: impact of timing of immunization information. Pediatrics. 2011 May;127 Suppl 1(Suppl 1):S120-6. doi: 10.1542/peds.2010-1722R. Epub 2011 Apr 18. PMID 21502250
- [Derived] Kriss JL, Frew PM, Cortes M, Malik FA, Chamberlain AT, Seib K, Flowers L, Ault KA, Howards PP, Orenstein WA, Omer SB. Evaluation of two vaccine education interventions to improve pertussis vaccination among pregnant African American women: A randomized controlled trial. Vaccine. 2017 Mar 13;35(11):1551-1558. doi: 10.1016/j.vaccine.2017.01.037. Epub 2017 Feb 16. PMID 28216190